CLINICAL TRIAL: NCT06086171
Title: Perioperative Methadone Compared to Placebo in Elderly Hip Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHS-An-4-2023
Record Dates: First submitted 2023-10-04; First posted 2023-10-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hip Fractures; Methadone
Keywords: Hip fractures; Elderly; Fragile; methadone; perioperative; analgesic treatment; pain; verbal rating scale; morphine consumption
MeSH Terms: conditions — Hip Fractures; Pain | interventions — Methadone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone (Experimental): Methadone hydrochloride (0.10 mg/kg) administered intravenously at the induction of anaesthesia
  Interventions: Drug: Methadone Hydrochloride
- Placebo (Placebo Comparator): Standard saline solution administered intravenously at the induction of anaesthesia
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methadone Hydrochloride — Methadone hydrochloride (0.10 mg/kg) administered intravenously at the induction of anaesthesia
  Other Names: Methadone
  Arms: Methadone
Other: Placebo — Saline solution
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Hip fractures are associated with severe pain and are sustained by the elderly population. Demand for adequate pain relief combined with a low tolerance for analgesic drugs makes the treatment of elderly hip fracture patients difficult. Perioperative methadone could improve the analgesic treatment of these patients. An earlier pilot study showed that 0.10 mg/kg was safe to use. This study further investigates the advantages of methadone. The study's objective is to investigate the analgesic effects of a single dose of methadone given during hip fracture surgery.

DETAILED DESCRIPTION:
Studies investigating the perioperative use of methadone have shown promising analgesic properties. Our pilot study (EudraCT no.: 2022-001857-22) showed that a dosage of 0.10 mg/kg was safe to use and showed excellent analgesic properties. Sufficient management of acute postoperative pain is important in relation to morbidity, hospital costs, and mortality. About 60% of patients undergoing surgical intervention experience moderate to severe postoperative pain. Thus, sufficient analgesic treatment is crucial in the initial postoperative days, which are considered the most painful phase of recovery. Opioids have conventionally been used as an analgesic treatment in this phase. However, this treatment has been accompanied by side effects and addiction. Methadone shares these side effects, however, as methadone only needs to be administered once, the risk of side effects decreases significantly. This study will investigate the analgesic effects of a single dose of methadone given during hip fracture surgery.

The first objective is to investigate the analgesic effect of perioperative methadone compared with a placebo in acute hip fracture surgery. The second objective is to investigate the long-term effects of methadone on continued opioid consumption, pain, and mobility three months after surgery.

The null hypothesis is that there is no difference in postoperative pain, opioid consumption, or related side effects if a patient receives a dose of methadone or placebo during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an acute hip fracture (incurred <24 hours ago) on x-rays in the emergency department (ED) at the university hospital of southern Denmark (SHS). This includes collum femoris fractures, pertrochanteric fractures, and subtrochanteric fractures.
* Patients must be able to read and understand Danish.

Exclusion Criteria:

* Multiple fractures or multi-trauma patient
* Previous allergic reactions or hypersensitivity towards methadone hydrochloride or sodium chloride
* Health conditions preventing treatment:

Chronic obstructive pulmonary disease with either past exacerbations or daily symptoms History of acute asthma attacks History of drug-induced eczema Pulmonary hypertension Raised intracranial pressure or recent head injury Pheochromocytoma History of paralytic ileus QT-interval prolongation on electrocardiogram (ECG) Myasthenia gravis Known liver disorder Hypotension (systolic blood pressure <100 mmHg at admission) Acute pancreatitis Severe kidney disease (GFR ≤10)

* Concurrent administration with MAO inhibitors or within 2 weeks of suspending treatment with these medicinal products
* Concurrent administration of benzodiazepines
* Impaired cognitive function e.g. dementia. Patients must be able to give informed consent and be able to ask for rescue analgesics if needed
* Current opioid addiction or intravenous addiction

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Consumption of daily morphine equivalents 3 days post operatively | 3 days post-surgery
  All opioids (short-acting and long-acting) will be converted into daily morphine milligram equivalent doses. The amount of opioids used by the patient within the last 24 hours will be registered daily. A minimum amount of 0 mg and a maximum amount of 150 mg can be recorded.
Consumption of daily morphine equivalents 3 months post operatively | 3 months post-surgery
  The opioid consumption will be registered as a mean daily consumption of both long-acting opioids and rescue medication prescribed in the medication chart and reported by the patient. Different types of opioids will be converted into the daily morphine milligram equivalent dose. Minimum score will be 0 mg and the maximum will be 150 mg.

SECONDARY OUTCOMES:
Postoperative pain assessment with verbal rating scale (VRS) | 3 days post-surgery
  Patients will be asked to assess pain intensity daily in the hip both at rest and when mobilized. Pain intensity will be evaluated using the verbal rating scale consisting of five choices - 1 (No pain), 2 (Slight pain), 3 (Moderate pain), 4 (Severe pain), and 5 (Unbearable pain).
Time until patient first stands up post-surgery | up to 72 hours post-surgery
  This will be registered in hours and minutes. The minimum is 0 hours and 0 minutes and the maximum is 72 hours and 0 minutes.
Mobility assessment using the Cumulated Ambulation Score (CAS) | 3 days post-surgery
  The cumulated ambulation score describes the patient's independence with regard to three activities. The first getting in and out of bed, the second ability to transition from sit-to-stand-to-sit from a chair, and the third is walking ability. Each of these activities is assessed on a three-point scale from 0-2 (0 = Not able to, despite human assistance and verbal cueing, 1 = Able to, with human assistance and/or verbal cueing from one or more persons, 2 = Able to safely, without human assistance or verbal cueing. A CAS score will range from zero (worst) to six (best) and will be measure daily.
Number of patients with post operative nausea or vomiting (PONV) | 3 days post-surgery
  Postoperative nausea or vomiting (PONV) will be registered binomial as "yes" or "no" once daily
Number of days to discharge after surgery | From admission to the ward to discharge, up to 14 days
  The number of days from ward admission until discharge. Patients moved to another department are still considered hospitalized. The minimum is 0 days and the maximum is 14 days.
Number of patients requiring an antidote | 3 days post-surgery
  Administration of an antidote will be registered binomial as "yes" or "no". Indications for the use of an antidote include a respiratory frequency of <10/min with peripheral oxygenation of <94% despite 4 liters of oxygen/minute, clinical signs of opioid overdose e.g. disproportionate drowsiness, or if the orthopaedic resident deems it necessary.
Number of patients with delirium assessed using the Confusion Assessment Method (CAM) | 3 days post-surgery
  Patients will be monitored using the confusion assessment method for signs of delirium. The method is binomial so that 0 means no signs of delirium and 1 means a patient is delirious.
Number of participants with constipation | 3 days post-surgery
  Occurrence of constipation during admission will be registered binomial as "yes" or "no". A patient with no bowel movements for ≥2 days is considered constipated.
Postoperative pain assessment with verbal rating scale (VRS) | 3 months post-surgery
  Patients will be asked to assess pain intensity daily in the hip both at rest and when mobilized. Pain intensity will be evaluated using the verbal rating scale consisting of five choices - 1 (No pain), 2 (Slight pain), 3 (Moderate pain), 4 (Severe pain), and 5 (Unbearable pain).
Quality of life assessed using EQ-5D-5L questionnaire | 3 months post-surgery
  The questionnaire comprises of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Patient mobility assessed using the new mobility score (NMS) | 3 months post-surgery
  New mobility score assesses gait; inside the home, outside the home and whilst shopping. A score of 0-3 points is given for each of these three functions, resulting in a total score between 0-9 points.
Number of persistent side effects | 3 months post-surgery
  The persistent presence of potential adverse reactions will be registered. This includes disproportional dizziness, vertigo, nausea, vomiting, constipation, and drowsiness.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Ougaard Schønnemann, Study Director — Sygehus Sønderjylland (Region Syddanmark)
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nygaard KH, Strom T, Specht K, Petersen SR, Schonnemann JO. Perioperative methadone compared to placebo in elderly hip fracture patients: a study protocol for a randomized controlled trial (MetaHip trial). Trials. 2024 Dec 20;25(1):842. doi: 10.1186/s13063-024-08694-6. PMID 39707407